CLINICAL TRIAL: NCT06686914
Title: The Effects of Cannabidiol on the Driving Performance of Healthy Adults by Dose and Sex
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Toni Marie Rudisill, Associate Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2311874160; 1R01DA058678-01A1 (NIH)
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Cannabidiol Effects; Driving Performance
MeSH Terms: interventions — Cannabidiol; Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cannabidiol (CBD) Oil 300mg (Active Comparator): Cannabidiol (CBD) Oil, 300mg, 1 dose, 120 minutes prior to testing. After consumption of the respective treatment drug, the participant will be given a standardized meal and wait for 120 minutes to allow for drug absorption and for CBD to begin taking effect; this time frame was chosen based on the pharmacokinetics of CBD along with the consideration of participant burden (max absorption 2-5 hours; average half-life 17 hours).
  Interventions: Drug: Cannabidiol (CBD) Oil 300mg
- Cannabidiol (CBD) Oil 150mg (Active Comparator): Cannabidiol (CBD) Oil, 150mg, 1 dose, 120 minutes prior to testing. After consumption of the respective treatment drug, the participant will be given a standardized meal and wait for 120 minutes to allow for drug absorption and for CBD to begin taking effect; this time frame was chosen based on the pharmacokinetics of CBD along with the consideration of participant burden (max absorption 2-5 hours; average half-life 17 hours).
  Interventions: Drug: Cannabidiol (CBD) Oil 150mg
- Placebo Oil (Placebo Comparator): Placebo Oil 1 dose 120 minutes prior to testing. After consumption of the respective treatment drug/placebo, the participant will be given a standardized meal and wait for 120 minutes to allow for drug absorption and for CBD to begin taking effect; this time frame was chosen based on the pharmacokinetics of CBD along with the consideration of participant burden (max absorption 2-5 hours; average half-life 17 hours).
  Interventions: Drug: Placebo Oil

INTERVENTIONS:
Drug: Cannabidiol (CBD) Oil 300mg — Cannabidiol (CBD) Oil 300mg, 1 dose
  Arms: Cannabidiol (CBD) Oil 300mg
Drug: Cannabidiol (CBD) Oil 150mg — Cannabidiol (CBD) Oil 150mg, 1 dose
  Arms: Cannabidiol (CBD) Oil 150mg
Drug: Placebo Oil — Placebo Oil, 1 dose
  Arms: Placebo Oil

SUMMARY:
The objectives/purpose of this study are to comprehensively investigate the effects of non-prescription CBD on driving performance, drowsiness, sedation, and cognitive function in a large sample of healthy adults aged 18-30 years, with additional characterization of effects by dose and by sex, using a rigorous RCT design which will naturally mitigate confounding factors.

ELIGIBILITY:
Inclusion Criteria:

* Possess a current drivers' license
* Driven a motor vehicle at least once in the past 30 days
* Able to read English
* Test negative for all substances on a urine drug test and complete a test drive to ensure the absence of simulation sickness
* Not taking any daily prescription medications (excluding birth control)
* Not diagnosed with any serious chronic disease by a licensed healthcare provider (including but not limited to Alzheimer's and related dementias, Parkinson's disease or other neurodegenerative disorder, major depressive or anxiety disorder, schizophrenia or other serious mental illness, arrhythmias, cataracts, glaucoma, chronic obstructive pulmonary disease, diabetes, epilepsy, sleep apnea, and fibromyalgia)
* Have an individual willing to drive them home after testing or be taken home by study staff after testing

Exclusion Criteria:

* Currently smoke, vape or use tobacco products, used CBD in the past 30 days
* Used illegal drugs in the past 30 days (e.g., cocaine/crack, heroin, methamphetamine, 3,4-methylenedioxy-methamphetamine, inhalants, phencyclidine, lysergic acid diethylamide, psilocybin mushrooms, or marijuana)
* Are pregnant or lactating at time of study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Mean standard deviation of lateral position | 150 minutes post intervention
  The driving simulator will measure mean standard deviation which is the amount a driver is weaving within the lane during the drive. Ranges from 0 to infinity, with higher means indicating worse performance.
Number of collisions | 150 minutes post intervention
  The driving simulator will measure how many times a participant crashes into other vehicles, signs, pedestrians, etc. during the simulation. Ranges from 0 to infinity, with higher numbers indicating worse performance.
Mean reaction time to stimuli | 150 minutes post intervention
  The driving simulator will measure the mean reaction time (seconds) that it takes for a person to brake when exposed to stimuli. Ranges from 0 to infinity, with higher means indicating worse performance.
Percent of time driver is out of travel lane | 150 minutes post intervention
  The driving simulator will measure the percent of time that each driver spends driving outside their travel lane. Percent ranges from 0-100, with higher scores indicating worse performance.

SECONDARY OUTCOMES:
Self-reported sleepiness scale | baseline
  Sleepiness will be assessed via the Stanford Sleepiness Scale which is a one question Likert scale question that ask a person's sleepiness level at that moment in time. The scale ranges from 1-7 with higher scores indicating more sleepiness. This test will be administered on a laptop.
Self-reported sleepiness scale | 200 minutes post intervention
  Sleepiness will be assessed via the Stanford Sleepiness Scale which is a one question Likert scale question that ask a person's sleepiness level at that moment in time. The scale ranges from 1-7 with higher scores indicating more sleepiness. This test will be administered on a laptop.
Mental sedation score | baseline
  The Visual Analog Mood Scale is a 16 question Likert type scale that assess different facets of a person's mental state. Questions 1,4,11, and 13 are summed together to get a mental sedation score. Higher scores indicate more sedation. This ranges from 0-400.This test will be administered on a laptop.
Mental sedation score | 200 minutes post intervention
  The Visual Analog Mood Scale is a 16 question Likert type scale that assess different facets of a person's mental state. Questions 1,4,11, and 13 are summed together to get a mental sedation score. Higher scores indicate more sedation. This ranges from 0-400.This test will be administered on a laptop.
Physical sedation score | baseline
  The Visual Analog Mood Scale is a 16 question Likert type scale that assess different facets of a person's mental state. Questions 3,5,6, and 16 are summed together to get a physical sedation score. Higher scores indicate more physical sedation. This ranges from 0-400. This test will be administered on a laptop.
Physical sedation score | 200 minutes post intervention
  The Visual Analog Mood Scale is a 16 question Likert type scale that assess different facets of a person's mental state. Questions 3,5,6, and 16 are summed together to get a physical sedation score. Higher scores indicate more physical sedation. This ranges from 0-400. This test will be administered on a laptop.
Mean reaction time to stimuli for PVT | baseline
  The psychomotor vigilance test is given via a computer program and assesses different facets of a person's vigilance, or ability to pay attention. It will measure a participants mean reaction time to the stimuli presented (in milliseconds). Higher times indicate worse performance. This ranges from 0 to infinity.
Mean reaction time to stimuli for PVT | 200 minutes post intervention
  The psychomotor vigilance test is given via a computer program and assesses different facets of a person's vigilance, or ability to pay attention. It will measure a participants mean reaction time to the stimuli presented (in milliseconds). Higher times indicate worse performance. This ranges from 0 to infinity.
Number of lapses in attention for PVT | Baseline
  The psychomotor vigilance test is given via a computer program and assesses different facets of a person's vigilance, or ability to pay attention. It will measure a participants number of lapses in attention to presented stimuli. The test considers any reaction over 500 milliseconds to be a lapse in attention. More lapses indicate worse performance. This ranges from 0 to infinity.
Number of lapses in attention for PVT | 200 minutes post intervention
  The psychomotor vigilance test is given via a computer program and assesses different facets of a person's vigilance, or ability to pay attention. It will measure a participants number of lapses in attention to presented stimuli. The test considers any reaction over 500 milliseconds to be a lapse in attention. More lapses indicate worse performance. This ranges from 0 to infinity.
Mean lapse duration for PVT | Baseline
  The psychomotor vigilance test is given via a computer program and assesses different facets of a person's vigilance, or ability to pay attention. It will measure a participants number of lapses in attention to presented stimuli. The test considers any reaction over 500 milliseconds to be a lapse in attention. It measures the mean lapse duration for each participant. Longer lapses indicate worse performance. This ranges from 0 to infinity.
Mean lapse duration for PVT | 200 minutes post intervention
  The psychomotor vigilance test is given via a computer program and assesses different facets of a person's vigilance, or ability to pay attention. It will measure a participants number of lapses in attention to presented stimuli. The test considers any reaction over 500 milliseconds to be a lapse in attention. It measures the mean lapse duration for each participant. Longer lapses indicate worse performance. This ranges from 0 to infinity.
Number of errors for PVT | Baseline
  The psychomotor vigilance test is given via a computer program and assesses different facets of a person's vigilance, or ability to pay attention. It will measure how many errors a person makes during the 10-minute test. More errors indicate worse performance. This ranges from 0 to infinity.
Number of errors for PVT | 200 minutes post intervention
  The psychomotor vigilance test is given via a computer program and assesses different facets of a person's vigilance, or ability to pay attention. It will measure how many errors a person makes during the 10-minute test. More errors indicate worse performance. This ranges from 0 to infinity.
Interference score for mean reaction on FT | Baseline
  The Flanker Task is administered on a laptop. The test assesses the mean reaction time to congruent and incongruent scenarios presented to participants. The score is the difference when subtracting the mean reaction time for congruent scenarios from the mean reaction time for incongruent scenarios. Larger differences indicate more impairment.
Interference score for mean reaction on FT | 200 minutes post intervention
  The Flanker Task is administered on a laptop. The test assesses the mean reaction time to congruent and incongruent scenarios presented to participants. The score is the difference when subtracting the mean reaction time for congruent scenarios from the mean reaction time for incongruent scenarios. Larger differences indicate more impairment.
Interference score for accuracy on FT | Baseline
  The Flanker Task is administered on a laptop. The test assesses the mean accuracy to congruent and incongruent scenarios presented to participants. The score is the difference when subtracting the mean accuracy for congruent scenarios from the mean accuracy for incongruent scenarios. Larger differences indicate more impairment.
Interference score for accuracy on FT | 200 minutes post intervention
  The Flanker Task is administered on a laptop. The test assesses the mean accuracy to congruent and incongruent scenarios presented to participants. The score is the difference when subtracting the mean accuracy for congruent scenarios from the mean accuracy for incongruent scenarios. Larger differences indicate more impairment.
Time to accurately complete the Trail Making Test Part A | Baseline
  Trail Making Test A provides an assessment of complex attention. This test is typically ended after 5 minutes. Thus, possible outcomes are 1-300 seconds. Greater time indicates more impairment.
Time to accurately complete the Trail Making Test Part A | 200 minutes post intervention
  Trail Making Test A provides an assessment of complex attention. This test is typically ended after 5 minutes. Thus, possible outcomes are 1-300 seconds. Greater time indicates more impairment.
Time to accurately complete the Trail Making Test Part B | Baseline
  TMT Part B is a neuropsychological test that assesses a person's ability to switch cognitive sets and process information. This test is typically ended after This test is typically ended after 5 minutes. thus, possible outcomes are 1-300 seconds. Greater time indicates more impairment.
Time to accurately complete the Trail Making Test Part B | 200 minutes post intervention
  TMT Part B is a neuropsychological test that assesses a person's ability to switch cognitive sets and process information. This test is typically ended after This test is typically ended after 5 minutes. thus, possible outcomes are 1-300 seconds. Greater time indicates more impairment.
Total recalled words on the Hopkins Verbal Learning test | Baseline
  The Hopkins Verbal Learning test assesses an individual's ability to learn a list of 12 words over 3 different learning trials. Ranges from 0 to infinity. Greater numbers of recalled words mean better performance.
Total recalled words on the Hopkins Verbal Learning test | 200 minutes post intervention
  The Hopkins Verbal Learning test assesses an individual's ability to learn a list of 12 words over 3 different learning trials. Ranges from 0 to infinity. Greater numbers of recalled words mean better performance.
Discrimination index for the Hopkins Verbal Learning test | Baseline
  The Hopkins Verbal Learning test assesses an individual's ability to learn a list of 12 words over 3 different learning trials. Ranges from 0 to infinity. The discrimination index is calculated by taking the number of hits minus the number of false positives. Higher values indicate better performance.
Discrimination index for the Hopkins Verbal Learning test | 200 minutes post intervention
  The Hopkins Verbal Learning test assesses an individual's ability to learn a list of 12 words over 3 different learning trials. Ranges from 0 to infinity. The discrimination index is calculated by taking the number of hits minus the number of false positives. Higher values indicate better performance.
Percentage correctness of response on Stroop Test | Baseline
  The Stroop Test is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute. Ranges from 0-100%. The higher the percentage, the more accurate.
Percentage correctness of response on Stroop Test | 200 minutes post intervention
  The Stroop Test is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute. Ranges from 0-100%. The higher the percentage, the more accurate.
Number congruent responses on Stroop Test | Baseline
  The Stroop Test is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute. Ranges from 0-infinity. Higher numbers indicate better performance.
Number congruent responses on Stroop Test | 200 minutes post intervention
  The Stroop Test is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute. Ranges from 0-infinity. Higher numbers indicate better performance.
Number incongruent responses on Stroop Test | Baseline
  The Stroop Test is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute. Ranges from 0-infinity. Higher numbers indicate worse performance
Number incongruent responses on Stroop Test | 200 minutes post intervention
  The Stroop Test is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute. Ranges from 0-infinity. Higher numbers indicate worse performance
Sum of scores for forward and backward responses on Digit Span test | Baseline
  The digit span test is a very short test that evaluates a person's cognitive status. It is frequently used in hospitals and physicians' offices in order for a clinician to quickly evaluate whether a person's cognitive abilities are normal or impaired. Ranges from 0 to infinity. Participant receives a score if they recall a numbered sequence in the forward and backward direction. If the sequence is correct, a point is earned. Higher scores indicate better performance.
Sum of scores for forward and backward responses on Digit Span test | 200 minutes post intervention
  The digit span test is a very short test that evaluates a person's cognitive status. It is frequently used in hospitals and physicians' offices in order for a clinician to quickly evaluate whether a person's cognitive abilities are normal or impaired. Ranges from 0 to infinity. Participant receives a score if they recall a numbered sequence in the forward and backward direction. If the sequence is correct, a point is earned. Higher scores indicate better performance.
Gestalt score based on correctness of clock drawing | Baseline
  The Clock Drawing Test (CDT) is a screening tool for cognitive impairment. Score ranges from 0-5. Higher scores indicate an accurate drawing.
Gestalt score based on correctness of clock drawing | 200 minutes post intervention
  The Clock Drawing Test (CDT) is a screening tool for cognitive impairment. Score ranges from 0-5. Higher scores indicate an accurate drawing.
Number of correct and non-duplicate responses on Animal Naming test | Baseline
  Animal Naming Test is a semantic fluency test that consists of listing as many names of animals as possible in 1 minute. Ranges from 0-infinity. The higher the number, the better the performance.
Number of correct and non-duplicate responses on Animal Naming test | 200 minutes post intervention
  Animal Naming Test is a semantic fluency test that consists of listing as many names of animals as possible in 1 minute. Ranges from 0-infinity. The higher the number, the better the performance.
Number of omission errors on N-back test | Baseline
  Ranges from 0-infinity. More errors indicate worse performance
Number of omission errors on N-back test | 200 minutes post intervention
  The n-back task is a continuous performance task that is commonly used as an assessment in psychology and cognitive neuroscience to measure a part of working memory and working memory capacity. The subject is presented with a sequence of stimuli, and the task consists of indicating when the current stimulus matches the one from n steps earlier in the sequence. Ranges from 0-infinity. More errors indicate worse performance
Number of commission errors on N-Back test | Baseline
  The n-back task is a continuous performance task that is commonly used as an assessment in psychology and cognitive neuroscience to measure a part of working memory and working memory capacity. The subject is presented with a sequence of stimuli, and the task consists of indicating when the current stimulus matches the one from n steps earlier in the sequence. Ranges from 0-infinity. More errors indicate worse performance
Number of commission errors on N-Back test | 200 minutes post intervention
  The n-back task is a continuous performance task that is commonly used as an assessment in psychology and cognitive neuroscience to measure a part of working memory and working memory capacity. The subject is presented with a sequence of stimuli, and the task consists of indicating when the current stimulus matches the one from n steps earlier in the sequence. Ranges from 0-infinity. More errors indicate worse performance
Percent correct matches on N-Back test | Baseline
  The n-back task is a continuous performance task that is commonly used as an assessment in psychology and cognitive neuroscience to measure a part of working memory and working memory capacity. The subject is presented with a sequence of stimuli, and the task consists of indicating when the current stimulus matches the one from n steps earlier in the sequence. Ranges from 0-100%. Higher percent correct is better performance
Percent correct matches on N-Back test | 200 minutes post intervention
  The n-back task is a continuous performance task that is commonly used as an assessment in psychology and cognitive neuroscience to measure a part of working memory and working memory capacity. The subject is presented with a sequence of stimuli, and the task consists of indicating when the current stimulus matches the one from n steps earlier in the sequence. Ranges from 0-100%. Higher percent correct is better performance

CONTACTS AND LOCATIONS:
Overall Officials: Toni M Rudisill, PhD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States